CLINICAL TRIAL: NCT03354325
Title: The Bronchiolitis Follow-up Intervention Trial
Acronym: BeneFIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Stanford University (Other)
Responsible Party: Principal Investigator, Eric Coon, MD, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 82296
Record Dates: First submitted 2017-11-15; First posted 2017-11-27 (Actual); Results first posted 2020-05-19 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Bronchiolitis
Keywords: Office Visits
MeSH Terms: conditions — Bronchiolitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Scheduled PCP follow-up (Active Comparator): Parents of children randomized to scheduled follow up will be instructed to follow up with their primary care physician (PCP) within 4 days of discharge regardless of improvement and/or symptom resolution. Research coordinators will verify that the child has a scheduled follow up appointment prior to discharge.
  Interventions: Behavioral: Scheduled PCP follow-up
- As needed PCP follow-up (Experimental): At the time of hospital discharge, parents will be instructed that the child does not need to automatically follow up with his/her primary care physician (PCP). Rather, the child should follow up on an as needed basis: if the child does not improve or if new concerns arise.
  Interventions: Behavioral: As needed PCP follow-up

INTERVENTIONS:
Behavioral: Scheduled PCP follow-up — Parents of children randomized to scheduled follow up will be instructed to follow up with their primary care physician within 4 days of discharge regardless of improvement and/or symptom resolution. Research coordinators will verify that the child has a scheduled follow up appointment prior to discharge.
  Arms: Scheduled PCP follow-up
Behavioral: As needed PCP follow-up — At the time of hospital discharge, parents will be instructed that the child does not need to automatically follow up with his/her primary care physician. Rather, the child should follow up on an as needed basis: if the child does not improve or if new concerns arise.
  Arms: As needed PCP follow-up

SUMMARY:
This study evaluates the value of routine follow-up with a child's pediatrician after hospitalization for bronchiolitis. Parents of half of participants will be instructed to follow-up with the child's pediatrician regardless of symptom resolution, while the other half will be instructed to follow-up on an as-needed basis (only if the child worsens, doesn't improve, or other concerns develop).

DETAILED DESCRIPTION:
Bronchiolitis is highly prevalent and burdensome among children less than 2 years of age. For this reason, many therapies have been tried by providers and studied by researchers. Unfortunately, interventions have largely been shown to be ineffective, prompting campaigns to reduce use of ineffective therapies. One commonly prescribed but thus far unstudied intervention often provided to children discharged after hospitalization for bronchiolitis is routine follow up with their pediatrician. Whether the costs and time spent for these visits are worthwhile depends on the extent to which the child and the child's parents benefit.

ELIGIBILITY:
Inclusion Criteria:

* Children less than two years of age who are hospitalized with an attending physician diagnosis of bronchiolitis.

Exclusion Criteria:

* Chronic lung disease
* Complex or hemodynamically significant heart disease
* Immunodeficiency
* Neuromuscular disease
* Discharged home with medication for withdrawal
* Inpatient team believes the child should follow up with their PCP

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 304 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-04-24 (Actual); Study Completion 2019-05-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Coon, MD, MS, Principal Investigator — University of Utah
Locations (4):
- United States (4):
  - Packard El Camino Hospital, Mountain View, California
  - Lucile Packard Children's Hospital, Palo Alto, California
  - Intermountain Riverton Hospital, Riverton, Utah
  - Primary Children's Hospital, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Ridd MJ, Lewis G, Peters TJ, Salisbury C. Patient-doctor depth-of-relationship scale: development and validation. Ann Fam Med. 2011 Nov-Dec;9(6):538-45. doi: 10.1370/afm.1322. PMID 22084265
- [Background] Thayaparan AJ, Mahdi E. The Patient Satisfaction Questionnaire Short Form (PSQ-18) as an adaptable, reliable, and validated tool for use in various settings. Med Educ Online. 2013 Jul 23;18:21747. doi: 10.3402/meo.v18i0.21747. No abstract available. PMID 23883565
- [Derived] Willer RJ, Brady PW, Tyler AN, Treasure JD, Coon ER. The Current State of High-Flow Nasal Cannula Protocols at Children's Hospitals. Hosp Pediatr. 2023 May 1;13(5):e109-e113. doi: 10.1542/hpeds.2022-006969. PMID 37051799
- [Derived] Coon ER, Schroeder AR, Lion KC, Ray KN. Disparities by Ethnicity in Enrollment of a Clinical Trial. Pediatrics. 2022 Feb 1;149(2):e2021052595. doi: 10.1542/peds.2021-052595. No abstract available. PMID 35043194
- [Derived] Coon ER, Hester G, Ralston SL. Why Are So Many Children With Bronchiolitis Going to the Intensive Care Unit? JAMA Pediatr. 2022 Mar 1;176(3):231-233. doi: 10.1001/jamapediatrics.2021.5186. No abstract available. PMID 34928316
- [Derived] Willer RJ, Johnson MD, Cipriano FA, Stone BL, Nkoy FL, Chaulk DC, Knochel ML, Kawai CK, Neiswender KL, Coon ER. Implementation of a Weight-Based High-Flow Nasal Cannula Protocol for Children With Bronchiolitis. Hosp Pediatr. 2021 Aug;11(8):891-895. doi: 10.1542/hpeds.2021-005814. Epub 2021 Jul 7. PMID 34234010
- [Derived] Chi KW, Coon ER, Destino L, Schroeder AR. Parental Perspectives on Continuous Pulse Oximetry Use in Bronchiolitis Hospitalizations. Pediatrics. 2020 Aug;146(2):e20200130. doi: 10.1542/peds.2020-0130. Epub 2020 Jul 16. PMID 32675334
- [Derived] Coon ER, Destino LA, Greene TH, Vukin E, Stoddard G, Schroeder AR. Comparison of As-Needed and Scheduled Posthospitalization Follow-up for Children Hospitalized for Bronchiolitis: The Bronchiolitis Follow-up Intervention Trial (BeneFIT) Randomized Clinical Trial. JAMA Pediatr. 2020 Sep 1;174(9):e201937. doi: 10.1001/jamapediatrics.2020.1937. Epub 2020 Sep 8. PMID 32628250

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Scheduled PCP Follow-up | As Needed PCP Follow-up
Started | 151 | 153
Completed | 131 | 138
Not Completed | 20 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Scheduled PCP Follow-up | As Needed PCP Follow-up | Total
Number analyzed (Participants) | 151 | 153 | 304
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 151 | 153 | 304
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 67 | 125
  Male | 93 | 86 | 179
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 34 | 56 | 90
  Not Hispanic or Latino | 117 | 97 | 214
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 11 | 12 | 23
  Native Hawaiian or Other Pacific Islander | 14 | 12 | 26
  Black or African American | 4 | 3 | 7
  White | 113 | 116 | 229
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 7 | 9 | 16

OUTCOME MEASURES:

1. Primary Outcome: Parental Anxiety
Description: Parental anxiety, as measured by the anxiety portion of the Hospital Anxiety and Depression Scale (HADS), a 0-28 point scale, with higher values representing higher anxiety.
Time Frame: Measured at the first data collection phone call (5-9 days following discharge).
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Scheduled PCP Follow-up | As Needed PCP Follow-up
Number analyzed (Participants) | 131 | 138
points on a scale | 4.2 (3.5) | 3.9 (3.5)

2. Secondary Outcome: Time From Hospital Discharge to Cough Resolution
Time Frame: Measured by parent report via weekly research coordinator phone calls, until symptoms resolved or 50 days after discharge, whichever occurs first.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Scheduled PCP Follow-up | As Needed PCP Follow-up
Number analyzed (Participants) | 131 | 138
days | 9.8 (8.2) | 9.2 (6.7)

3. Secondary Outcome: Time From Hospital Discharge to Child Reported Back to Normal
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Scheduled PCP Follow-up | As Needed PCP Follow-up
Number analyzed (Participants) | 131 | 138
days | 9.6 (8.7) | 8.8 (6.8)

4. Secondary Outcome: Number of Clinic Visits Prior to Symptom Resolution
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: visits
Arm/Group | Scheduled PCP Follow-up | As Needed PCP Follow-up
Number analyzed (Participants) | 131 | 138
visits | 1.1 (0.7) | 0.5 (0.7)

5. Secondary Outcome: Any Hospital Re-admission Prior to Symptom Resolution
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Scheduled PCP Follow-up | As Needed PCP Follow-up
Number analyzed (Participants) | 131 | 138
percent | 3.8 (1.9) | 2.2 (1.4)

6. Secondary Outcome: Any ED Visit Prior to Symptom Resolution
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Scheduled PCP Follow-up | As Needed PCP Follow-up
Number analyzed (Participants) | 131 | 138
percent | 3.8 (1.9) | 5.8 (2.3)

7. Secondary Outcome: Number of Missed Work Days
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Scheduled PCP Follow-up | As Needed PCP Follow-up
Number analyzed (Participants) | 131 | 138
days | 2.1 (4.1) | 1.6 (3.2)

8. Secondary Outcome: Missed Daycare
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Scheduled PCP Follow-up | As Needed PCP Follow-up
Number analyzed (Participants) | 131 | 138
days | 1.2 (3.5) | 0.8 (2.9)

9. Secondary Outcome: Ambulatory Prescriptions (Albuterol, Antibiotics, Steroids)
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Scheduled PCP Follow-up | As Needed PCP Follow-up
Number analyzed (Participants) | 131 | 138
percent | 16.0 (3.7) | 9.4 (2.9)

10. Secondary Outcome: Ambulatory Testing (i.e. Pulse Oximetry, Chest X-ray)
Time Frame: Measured by parent report, at the first data collection phone call (5-9 days following discharge).
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Scheduled PCP Follow-up | As Needed PCP Follow-up
Number analyzed (Participants) | 131 | 138
percent | 67 (47) | 22 (42)

11. Secondary Outcome: Relationship With PCP
Description: Measured by the Patient-Doctor Depth-of-Relationship Scale, 0-32 points, with higher scores indicating a stronger relationship with PCP.
Time Frame: Measured by parent report via research coordinator phone call at 1 month from discharge.
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Scheduled PCP Follow-up | As Needed PCP Follow-up
Number analyzed (Participants) | 131 | 138
points on a scale | 26.0 (6.3) | 26.5 (6.4)

12. Secondary Outcome: Report That Care Was Perfect 1 Month After Discharge
Description: Measured by a question from the Patient Satisfaction Questionnaire Short Form (PSQ-18), those who indicate agree or strongly agree
Time Frame: Measured by parent report via research coordinator phone call at 1 month from discharge.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Scheduled PCP Follow-up | As Needed PCP Follow-up
Number analyzed (Participants) | 116 | 128
percent | 99.2 (9.3) | 97.6 (15.2)

13. Secondary Outcome: Immunizations Received 1 Month After Discharge
Time Frame: Measured by parent report via research coordinator phone call at 1 month from discharge.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Scheduled PCP Follow-up | As Needed PCP Follow-up
Number analyzed (Participants) | 116 | 128
percent | 36.2 (48.3) | 32.8 (47.1)

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Scheduled PCP Follow-up | As Needed PCP Follow-up
All-Cause Mortality (participants affected / at risk) | 0/151 | 0/153
Serious Adverse Events (participants affected / at risk) | 0/151 | 0/153
Other Adverse Events (participants affected / at risk) | 0/151 | 0/153

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-01): https://cdn.clinicaltrials.gov/large-docs/25/NCT03354325/Prot_SAP_000.pdf